CLINICAL TRIAL: NCT07115004
Title: A Prospective, Multicenter, Open-label, Phase 3 Clinical Study to Evaluate the Efficacy and Safety of Prophylactic VGA039 in Adolescent and Adult Patients With Von Willebrand Disease (VIVID-6)
Brief Title: Study to Evaluate Subcutaneous (SC) VGA039 in Patients With Von Willebrand Disease (VWD)
Acronym: VIVID-6
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vega Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VGA039-CP002
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Von Willebrand Disease (VWD)
Keywords: VWD; von Willebrand Disease; VIVID-6; Vega Therapeutics; Star Therapeutics; VGA039
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Intervention Model Description: The study includes two sequential phases: an initial observational period, during which participants are monitored without receiving study drug, followed by an interventional period where eligible participants are assigned to receive the investigational product VGA039 for approximately 49 weeks. The interventional phase follows a single-group assignment model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Multiple Doses of VGA039 after observational run-in (Experimental): Participants who meet eligibility criteria and complete a 24-week observational phase will receive VGA039 SC for approximately 49 weeks.
  Interventions: Drug: VGA039

INTERVENTIONS:
Drug: VGA039 — VGA039 SC administered for 49-weeks during the interventional phase following a 24-week observational period.

SUMMARY:
This is a phase 3 study that will evaluate subcutaneous (SC) VGA039 in patients with von Willebrand Disease (VWD)

DETAILED DESCRIPTION:
This Phase 3 multicenter, open-label, single-sequence cross-over study will investigate the safety and efficacy of subcutaneous administration of VGA039 as prophylaxis for bleeding in patients with every type of VWD. The study consists of an Observational Period of at least 24 weeks followed by an Active Treatment Period of approximately 49 weeks of VGA039 treatment. Bleeding data and details of treatments used will be collected from each patient during both study periods. The number, duration, location, and types of bleeds experienced, as well as treatments for bleeds, will be recorded in patient diaries. Adverse events will also be monitored and recorded throughout both study periods.

ELIGIBILITY:
Key Inclusion Criteria

* 12 to 75 years of age, inclusive
* No clinically significant laboratory, ECG, or vital signs results
* Documented diagnosis consistent with VWD of any type
* Historical annualized bleeding rate (ABR; excluding menstrual bleeds and bleeds under the skin) of both untreated and treated bleeds ≥12 per year
* Patients with VWD who are judged by the investigator to be suitable candidates for routine prophylaxis to reduce the frequency of bleeding episodes
* Hemoglobin level ≥ 8 g/dL and platelet count ≥ 100 x 109/L at Screening

Key Exclusion Criteria

* Use of routine prophylaxis of VWF-containing concentrates defined as at least 1 VWF-containing concentrate infusion to prevent or reduce bleeding per week during the previous 6 months prior to screening
* Planning to initiate routine prophylaxis with VWF-containing concentrates or any other hemostatic treatment during the study
* Patients with pro-thrombotic disorders or abnormal findings on laboratory thrombophilia evaluation performed at screening or previously documented
* History of arterial or venous thrombosis, including superficial thrombophlebitis, or embolism
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular disease, cerebrovascular disease, peripheral vascular disease, or metabolic dysfunction
* Baseline FVIII activity > lower limit of normal (LLN)

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of bleeding events [Efficacy] | Time Frame: From 7 days after informed consent until 49 weeks after SC study drug initiation

SECONDARY OUTCOMES:
Incidence of treated bleeding events [Efficacy] | From 7 days from Informed consent until 49 weeks after SC study drug initiation
Incidence, nature and severity of adverse events (AEs) and serious adverse events (SAEs), including hypersensitivity, anaphylaxis, or anaphylactoid reactions | From informed consent until 49 weeks after SC study drug initiation
Plasma concentrations of SC doses of VGA039 | From just prior to the start of study drug administration until 49 weeks after SC study drug initiation
Incidence of Anti-drug antibodies to VGA039 | From just prior to the start of study drug administration until 49 weeks after SC study drug initiation

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Science 37, Inc. (Virtual Clinical MetaSite), Morrisville, North Carolina
  - Hemophilia Center of Western PA, Pittsburgh, Pennsylvania
  - Washington Center for Bleeding Disorders, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to legal, ethical, or regulatory restrictions related to the study population or data use agreements.